CLINICAL TRIAL: NCT01845922
Title: The Prevention of Refeeding Syndrome by a Diet Regime in Patient With Head and Neck Cancer
Brief Title: The Effect of a Diet Based on Low Sodium and Slowly Absorbed Carbohydrates on the Incidence of Refeeding Syndrome in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HKM refeeding
Record Dates: First submitted 2013-04-22; First posted 2013-05-03 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Refeeding Syndrome
Keywords: Refeeding Syndrome; low sodium; slowly absorbed carbohydrates; hypopotassemia; hypophosphatemia
MeSH Terms: conditions — Refeeding Syndrome; Hypokalemia; Hypophosphatemia | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low sodium diet (Experimental): Low sodium diet
  Interventions: Dietary Supplement: Low sodium diet
- Control (No Intervention): Standard diet regime

INTERVENTIONS:
Dietary Supplement: Low sodium diet — Low sodium diet
  Arms: Low sodium diet

SUMMARY:
The study is based on a master thesis which showed that 72% of patients with head and neck cancer admitted to a Danish hospital (Rigshospitalet, Copenhagen) developed refeeding syndrome after admission.

Refeeding syndrome is characterized by a decrease in plasma phosphate levels, which develops after the reintroduction of an adequate food intake after a longer period of starvation or semi-starvation. This normally happens within 7 days after reintroduction of food.

The aim of this study is to minimize the incidence of refeeding syndrome in this group of patients by reintroducing food slowly and by providing a diet low in sodium and high in slowly absorbed carbohydrates as a prevention diet (i.e. given before a potential decrease in plasma phosphate levels appear). Both patients that eat normally, patients with eating tubes and patients with central vein catheters are included in the study, but the data will be evaluated both together and separately.

DETAILED DESCRIPTION:
A large weight loss as a result of a longer period (>30 days) of starvation or semi-starvation will result in a metabolic adaptation to the decreased food intake. To prevent the degradation of muscle mass into gluco- and ketogenic amino acids to be used for energy production, a shift from gluconeogenesis to lipolysis occurs. Lipids therefore become the primary energy fuel, and the body adapts to use ketone bodies instead of glucose. The reduction in glucose metabolism results in a decreased need for amino acids for use in gluconeogenesis. This means that less amino acids are needed for gluconeogenesis and therefore important muscle mass is preserved. At the same time as the lipid stores are degraded, an intracellular depletion of phosphate, potassium and magnesium occurs. The serum levels of these electrolytes stay within the normal range as long as the body is in the adaptive starvation state. A too quick reintroduction of food to the body will result in a major glucose-induced increase in insulin secretion that will stimulate the transport of glucose, phosphate, potassium and magnesium from plasma into the cells. Because the extracellular blood volume is much smaller than the intracellular, an influx of these electrolytes to the intracellular space will result in a quick and large decrease in the plasma levels. Likewise, an influx of glucose means that it again can enter the glucolysis, and the need for phosphate and the co-factor thiamine, for the production of ATP, will increase. The increased production of adenosine triphosphate (ATP) will activate membrane pumps and reestablish the membrane potential. This means that sodium will be transported from the large intracellular space to the small extracellular, with subsequent fluid retention and edema formation.

Therefore a slowly introduced diet low in sodium and high in slowly absorbed carbohydrates might prevent the development of refeeding syndrome.

ELIGIBILITY:
Inclusion Criteria:

* authoritative
* written consent
* suspected of or diagnosed with head and neck cancer
* Increased risk of Refeeding syndrome, defined by one of the below:
* A-score of 1 in the Nutritional Risk Screening 2002 (NRS 2002)
* high levels of alcohol consumption (men>168g alcohol/week corresponding to approximately 14 units, women>84g alcohol/week corresponding to approximately 7 units)
* anamnesis with prior radiation therapy
* Head and neck pain that require pain management or inhibits food intake
* the presence of problems with eating that are so serious that the food intake is inhibited

Exclusion Criteria:

* minor or declared incapable of managing own affairs
* patients that are incapable of understanding and communicating in Danish
* patients with dementia
* if the patient is not diagnosed with head and neck cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Occurence of Refeeding events | daily, starting from day of admission and until day 7 of the treatment period or until discharge from the hospital if before day 7
  Measured by a decrease in plasma phosphate levels.

SECONDARY OUTCOMES:
Incidence of infections | daily, starting from day of admission and until day 7 of the treatment period or until discharge from the hospital if before day 7
  Measured by infection events recorded in the medical journal.
Length of stay | Number of days from admission until discharge from the hospital, assessed up to 6 month
  Measured by number of days in the hospital
Amount of days admitted to a Intensive-care unit | Number of days from admission until discharge from the Intensive-care unit, assessed up to 6 month
  Measured by number of days in the intensive-care unit
Other complications than infections | daily, starting from day of admission and until day 7 of the treatment period or until discharge from the hospital if before day 7
  Measured by thrombosis events and other complications recorded in the medical journal

OTHER OUTCOMES:
Nutritional status | daily, starting from day of admission and until day 7 of the treatment period or until discharge from the hospital if before day 7
  Measured by changes in plasma cobalamin levels/vitamin B12 levels (pmol/L), plasma iron levels (μmol/L), plasma ferritin levels (μg/L), mean cell volume (MCV) (fL), plasma albumin levels (μmol/L), plasma alanine aminotransferase levels (ALAT) (U/L), plasma coagulation factors II, VII, X levels (INR), plasma c-reactive protein levels (nmol/L), hemoglobin levels (Hgb) (mmol/L), plasma sodium levels (mmol/L), plasma potassium levels (mmol/L), plasma creatinine levels (μmol/L), plasma carbamide levels (mmol/L), plasma folate levels (nmol/L), plasma zink levels (μmol/L), plasma magnesium levels (mmol/L) and plasma selenium levels (μg/L).

CONTACTS AND LOCATIONS:
Overall Officials: Jens R. Andersen, MD, lektor, Principal Investigator — University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen Ø, Denmark